CLINICAL TRIAL: NCT06632249
Title: Effects of HIIT VR Exergame on Attention and Executive Function in Young People With ADHD: A Randomized Clinical Trial With 'Move Sapiens®'
Brief Title: Effects of HIIT VR Exergame on Attention and Executive Function in Young People With ADHD
Acronym: VRADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: University of Sao Paulo (Other); Centro de Inovação em Saúde Mental (CISM) (Unknown); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Grupo UniEDUK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-0540
Record Dates: First submitted 2024-09-30; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Virtual Reality (VR); High-Intensity Interval Training (HIIT)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: This study will be a single-blind clinical trial; the evaluators of the primary outcomes will be blinded, unaware of the group allocation to ensure the objectivity of the assessments. The data analysis will remain blinded to ensure that the researcher in charge is unaware of the experimental conditions, thus maintaining the impartiality of the analysis. However, the participants will be aware of their allocation group, as they will experience the different versions of the VR game 'Move Sapiens®'; one group will perform the exergame, with HIIT physical exercise, while the other will participate using a joystick, without physical exercise, which will prevent blinding of the volunteers. The training monitoring team, due to operational necessity, will also not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT VR (Experimental): The virtual reality (VR) exergame 'Move Sapiens®' will be implemented through the VR headset Oculus Quest 2 (Meta®, Menlo Park, USA). The game's objective is to take as much life from the drone as possible while avoiding being hit to preserve their own life, the drone not only moves erratically but also can attack, having a defined amount of life, just like the player. Participants will use a virtual exoskeleton to interact with the environment, and their main task is to aim and punch a drone that moves unpredictably. The exergame incorporates a short HIIT model, consisting of 12 cycles that include 16 seconds of maximum effort followed by 20 seconds of rest. This structured format is intrinsic to the game's design, aiming for a balance between effort and recovery. Essential factors for the simulation design include an engaging sensory experience of enhanced physical skills and the application of powerful punches in the game design.
  Interventions: Other: Practice with the virtual reality game
- Sedentary VR (Sham Comparator): Participants will play an adapted version of the 'Move Sapiens®' exergame in VR, which maintains the immersive environment of the original game but excludes any physical exercise component. In this version, interaction will be carried out exclusively through joystick manipulation, without requiring physical activity from the participants.
  Interventions: Other: Practice with the virtual reality game

INTERVENTIONS:
Other: Practice with the virtual reality game — 4 weeks of practice with the virtual reality game, totalling 20 sessions, 5 supervised in the laboratory and 15 at home with remote monitoring.
  Other Names: Move Sapiens®

SUMMARY:
The goal of this clinical trial is to learn if the "Move Sapiens" exergame in Virtual Reality (VR), incorporated with a short model of High-Intensity Interval Training (HIIT), works as an intervention tool for adolescents with Attention-Deficit Hyperactivity/Disorder (ADHD). It will also assess the safety and effectiveness of this intervention.

The main questions it aims to answer are: Does interacting with HIIT "Move Sapiens®" in VR improve attention and executive function in adolescents with ADHD? Does this intervention reduce other symptoms such as sleep problems and anxiety? Researchers will compare the HIIT VR exergame to a control condition.

Participants will: Engage with "Move Sapiens®" in VR (intervention group) or participate in a control condition with an adapted version of the exergame without physical exercise (control group) (five times a week for 4 weeks). Visit the clinic for assessments and tests. The analysis will involve comparing group means using a mixed model and calculating effect sizes with Cohen's d to determine the clinical relevance of the results

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) is a neurodevelopmental disorder characterized by inattention, hyperactivity, and impulsivity, affecting 3-5% of the global school-age population. Literature data show that high-intensity interval training (HIIT) is a potential intervention for ADHD inattentive symptoms and cognitive functioning deficits. These neuromodulatory effects have great potential to enhance neural plasticity and improve the executive functions of patients with ADHD. Furthermore, virtual reality (VR) can increase motivation for general activities, being a possible interesting tool, especially for people with ADHD.

Therefore, this study will investigate the potential of the 'Move Sapiens®' exergame in VR as an intervention tool for adolescents with ADHD. The primary objective is to assess whether interacting with 'Move Sapiens®' in VR can induce observable improvements in executive function and attention, a secondary objective is investigating a possible reduction in symptoms such as sleep problems and anxiety. Data will be obtained through validated questionnaires, in evaluation sessions conducted by clinicians and neuropsychologist, before and after the intervention. Ninety-eight participants, aged 12 to 17 with ADHD, will be randomly allocated in two groups that will interact with two versions of the VR 'Move Sapiens®' (with and without HIIT) during 20 sessions over 4 weeks. The four initial sessions and the last session will be performed in the laboratory. In these sessions, heart hate will also be monitored. Other sessions will be done at home with remote supervision. In all sessions, the game score will be monitored. The experimental group will practice the exergame, which incorporates a short model of HIIT, consisting of 12 cycles that include 16 seconds of maximum effort followed by 20 seconds of rest (total: 7 minutes and 12 seconds). In the control group, participants will engage in an adapted version of the Move Sapiens exergame without physical exercise, interacting through the joystick. This randomized clinical trial will be conducted in two centres: the Hospital de Clínicas de Porto Alegre (HCPA), and the Centro de Escola de Especialidades Médicas (CEEM - UniEduk/UniMax).

Furthermore, in a small convenience subsample of 30 participants (15 intervention and 15 control group) from the Porto Alegre-RS, we will explore a possible biological mechanism ("brain signature") associated with improved attention, detectable by fMRI, suggesting potential changes in brain function detectable through neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

* participants with diagnosis of ADHD according to DSM-5;
* age between 12 and 17 years;
* no prior use of ADHD medication or have not been using ADHD medication for at least one month.

Exclusion Criteria:

* participants with conditions and comorbidities that prevent the execution of HIIT in VR, such as severe additional psychiatric and physical conditions and a history of seizures;
* inattention score below 12 on the SNAP-IV inattention subscale;
* IQ below 70;
* recreationally active people who engage in intense, systematic physical activity more than two times a week.

For the MRI assessment, the following exclusionary criteria are added:

* participants with non-compatible aneurysm clips, cochlear implants, pacemakers, metal fragments in the body or eyes, or non-removable piercings;
* internal metal residues that interfere with image acquisition and analysis;
* severe claustrophobia;
* respiratory difficulties that prevent cooperation;
* inability to remain still due to hyperactivity;
* body weight and size exceeding device limits;
* excessive involuntary movement;
* anatomical abnormalities.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Inattention total score | Pre intervention (baseline) and post intervention (4th week)
  SNAP-IV will be used to assess inattention scores. Responses to 9 items aligned with DSM-5 Inatention criteria will be collected from parents using a 4-point Likert scale.
Inhibibitory Control | Pre intervention (baseline) and post intervention (4th week)
  Inhibitory control will be assessed with a computerized Go/No Go task. Number of Comission Errors corrected by age will be the outcome used.

SECONDARY OUTCOMES:
Verbal Working Memory | Pre intervention (baseline) and post intervention (4th week)
  The Digit Symbol Test evaluates verbal working memory and the outcome will be the scaled score for the backward condition.
Spatial Working Memory | Pre intervention (baseline) and post intervention (4th week)
  The Spatial Span Task is designed based on the Corsi Block, it evaluates spatial working memory. The outcome is the number of correct responses corrected by age for the backward condition
Cognitive Flexibility | Pre intervention (baseline) and post intervention (4th week)
  Trail Making Test will be used to evaluate cognitive flexibility. The outcome will be the time to complete B form corrected by age.
Reaction Time | Pre intervention (baseline) and post intervention (4th week)
  The Two-Choice Reaction Time task assesses processing speed and the score used will be the average reaction time corrected by age.
Sleep quality | Pre intervention (baseline) and post intervention (4th week)
  To assess sleep quality, we will use the Pittsburgh Sleep Quality Index (PSQI). This instrument is a self-administered questionnaire that investigates sleep quality over a one-month interval. The PSQI focuses on seven components: sleep latency, duration, efficiency, disturbances, use of sleep medication, daytime dysfunction, and subjective sleep quality. A higher total score on the PSQI indicates poorer sleep quality.
Anxiety symptoms | Pre intervention (baseline) and post intervention (4th week)
  To assess anxiety symptoms, we will use the 7-item Generalized Anxiety Disorder Scale (GAD-7). Participants will report the frequency of their anxiety symptoms over the past two weeks using a 4-point Likert scale, aiding in identifying and assessing the severity of generalized anxiety disorder.
Impulsivity and attention | Pre intervention (baseline) and post intervention (4th week)
  The MOXO-continuous performance test measures four domains, including attention, timeliness, hyperactivity and impulsivity. We will use the Impulsivity z-score to assess impulsivity.

OTHER OUTCOMES:
Functional Magnetic Resonance Imaging (fMRI) | Pre intervention (baseline) and post intervention (4th week)
  In a small convenience subsample from the Porto Alegre-RS group, fifteen participants from the intervention group and fifteen participants from the control group who provide informed consent (ICF) will have functional neuroimaging collected at the Brain Institute (InsCer) of PUCRS at baseline (T0) before the intervention, and within 7 days after the interventions (T1). The image acquisition time will be 40 minutes, and both resting-state fMRI and task-based fMRI images will be collected, using attention and inhibitory control tasks.
Heart Rate | Pre intervention (baseline) and post intervention (4th week)
  Heart rate (HR) data will be used as an objective measure of exercise intensity. HR recording will be evaluated during the 5 in-person training sessions, measuring the average and maximum HR (average HR and HRmax). A heart rate monitor (Polar H10) will be used for this purpose. Heart rate recovery (HRR: Δ bpm) will be measured during 5 minutes of recovery, and the average will be calculated every 5 seconds. Heart rate variability (HRV) will also be recorded (Polar beat app) and analysed using the Kubios software, in rest state and during a cognitive task.
Participants' experiences in the game | Pre intervention (baseline) and post intervention (4th week)
  The Game Experience Questionnaire will explore participants 'experiences related to the game, covering dimensions such as immersion, flow, and affect.
Discomfort associated with the use of virtual reality | Pre intervention (baseline) and post intervention (4th week)
  To assess discomfort associated with the use of virtual reality in our project, we will use the Simulator Sickness Questionnaire (SSQ). The 16-item questionnaire measures the incidence and severity of motion sickness symptoms in three categories: nausea, oculomotor issues, and disorientation.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Augusto Rohde, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (2):
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - UniEDUK-UniMax, Indaiatuba, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided